CLINICAL TRIAL: NCT05758805
Title: Esophageal Injury of a Tip CF Sensing Ablation Catheter for HP-SD of Paroxysmal and Persistent AF
Brief Title: Esophageal Injury of a Tip CF Sensing Ablation Catheter for HP-SD of Paroxysmal and Persistent AF (ESO-SAFE-HP-RF)
Acronym: ESO-SAFE-HP-RF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quovadis Associazione (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ESO-SAFE-HP-RF Study
Record Dates: First submitted 2023-02-21; First posted 2023-03-07 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation; Esophageal Perforation; Esophageal Fistula
Keywords: esophageal thermal injury (ETI); AF ablation; high-power, short-duration (HP-SD); mini-invasive esophagoscopy
MeSH Terms: conditions — Atrial Fibrillation; Esophageal Perforation; Esophageal Fistula

STUDY DESIGN:
Intervention Model Description: Pilot, about the safety, prospective, monocentric
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Unique Arm (Experimental): patients with atrial fibrillation and indication for radiofrequency ablation guided by electro-anatomical mapping with high-density mapping catheter and radiofrequency ablation by contact force ablation catheter, according to current guidelines
  Interventions: Device: mini-invasive esophagoscopy; Device: HP-SD AF ablation by a CF sensing catheter

INTERVENTIONS:
Device: mini-invasive esophagoscopy — mini-invasive esophagoscopy assessment of esophageal thermal injury (ETI) after an AF ablation session in an HP-SD setting, and with a tip CF sensing ablation catheter
Device: HP-SD AF ablation by a CF sensing catheter — AF ablation session in an HP-SD setting and with a tip CF sensing ablation catheter

SUMMARY:
This pilot, prospective, interventional, monocentric, independent, and no-profit clinical trial aims to investigate and evaluate the proportion, acute and chronic characteristics, and outcomes of esophageal thermal injury (ETI) in AF ablation using a high-power, short-duration (HP-SD) setting with contact force (CF) sensing tip ablation catheter in standard clinical practice. The main questions it aims to answer are:

* Evaluate the acute proportion of the ETI assessed by the mini-invasive esophagoscopy pre and post-procedure. In addition, clinical evaluations at 3, 6, and 12 months from the procedure are foreseen.
* Evaluate the contribution of the factors influencing RF procedure (contact force, impedance, RF power, RF time) on ETI development.
* Describe the relationship between the esophageal temperature (continuous monitoring) and ETI development.

DETAILED DESCRIPTION:
This study aims to estimate the proportion of esophageal thermal injury (ETI) as a result of the AF ablation using a high-power, short-duration (HP-SD) setting with contact force (CF) sensing tip ablation catheter immediately after and at 3, 6, and 12 months from the procedure, as well as describe their characteristics.

To be more sensitive and specific in detecting the presence of potentially chronic and progressing ETIs in esophageal ulcers and atrium-esophageal fistula, a minimally invasive esophagogastroscope will be used before (1-7 days) and after (1-3 days) the ablation procedure, with an internal comparison of the lesions observed. In addition, various clinical characteristics of the patients and descriptors of the ablation procedure (such as contact force, impedance, RF power, RF time, esophageal temperature, procedure times, etc.) will be collected and related to the presence of ETI.

The principal Medical Devices that will be used:

1. Cardiac Mapping system Ensite X (Abbott Medical),
2. Tip CF sensing catheter TactiFlex (Abbott Medical),
3. High mapping density catheter (HD GRID/Advisor FL, Abbott Medical),
4. Continuous temperature monitoring devices (Esotest Multi/Esotherm 7 poles, FIAB),
5. Video-endoscope EXERA III HDTV dual focus GIF-HQ190 (Olympus).

ELIGIBILITY:
Inclusion Criteria:

1. Atrial fibrillation and, according to current guidelines, indication for radiofrequency ablation guided by electro-anatomical mapping with high-density mapping catheter and radiofrequency ablation by contact force ablation catheter.
2. Able to sign the consent form.

Exclusion Criteria:

1. LVEF < 45%
2. Presence of thrombus in the left atrium
3. NYHA III/IV Class
4. Atrial diameter > 50mm
5. Moderate or severe valve dysfunction
6. Implanted ICD/CRT-D
7. Life expectancy < 1 year
8. Uncontrolled Hyperthyroidism
9. Hypertrophic or dilatative cardiomyopathy
10. Kidney failure (eGFR < 30)
11. Body Mass Index (BMI)> or = 35
12. Participation in another clinical trial in the past 3 months
13. Inability to express informed consent for the study
14. Patients with esophageal pathologies and a history of gastritis
15. Pregnancy (ascertained by performing the HCG test), breastfeeding, pregnancy planned during the study, or fertile female subjects who refused to use a highly effective contraceptive measure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of the acute esophageal thermal injury (ETI) | 1-3 days after AF ablation procedure
  Evaluate the acute proportion of the esophageal thermal injury (ETI)

SECONDARY OUTCOMES:
Factors influencing RF procedure on ETI development | 1-3 days after AF ablation procedure
  Contribution of the factors influencing RF procedure (contact force, impedance, RF power, RF time) on ETI development
Esophageal temperature by an esophageal continuous monitoring device | during AF ablation procedure
  Celsius degree.
ETI monitoring | 12 months after AF ablation procedure
  Chronic (every 3 months until healing) evaluation of discovered ETI.
AF ablation procedure times | 1 day
  minutes
AF recurrences | 12 months after AF ablation procedure
  AF recurrences until 12 months after the ablation procedure
Serious and no serious adverse events | 12 months after AF ablation procedure
  Serious and no serious adverse events after the ablation procedure

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Dello Russo, MD, Principal Investigator — Cardiology and Arrhythmology Dept., Azienda Ospedaliero Universitaria delle Marche, Ancona (Italy)
Locations (1):
- SOD di Cardiologia e Aritmologia, Ancona, Italy

IPD SHARING:
Plan to Share IPD: No
no IPD share planned